CLINICAL TRIAL: NCT03034993
Title: Improving Self-Management of Chronic Conditions Among Homeless Persons: a Community-Based Participatory Approach Using Text Messaging
Brief Title: Self-Management Using Text Messaging in a Homeless Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Boston Health Care for the Homeless Program (Unknown)
Responsible Party: Principal Investigator, Donald Keith McInnes, Research Assistant Professor, BUSPH, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-35967; catalyst grant (Other: BU SPH)
Record Dates: First submitted 2017-01-26; First posted 2017-01-27 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Chronic Disease
Keywords: Healthcare for homeless; Text messages; Primary care visits; Medication adherence; Inpatient admissions
MeSH Terms: conditions — Chronic Disease; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Messaging (Experimental): This group will receive text messages with appointment reminders, medication taking education and motivation, and for reporting of mood.
  Interventions: Behavioral: Text Messaging
- Control (Placebo Comparator): This group will receive simple text messages about general health promotion, such as about the importance of drinking water on hot days, using sunscreen, etc.
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Text Messaging — Subjects will receive text messages with reminders of their upcoming outpatient health care appointments at the Boston Health Care for the Homeless Program (BHCHP) clinic. The text message will indicate the time of the appointment and the location (e.g. "Remember appointment Friday March 15 at 10am in the Yawkey building"). Appointment reminder text messages will be sent 3 days ahead and again 1 day ahead of the appointment date. Medication related texts will be sent every other day and will be educational and motivational (e.g. "Keep taking medications that way the doctor prescribed them, even if feeling fine"). Mood related texts will also be sent every other day and ask about mood on a 1 to 5 scale. The participant will text back a response.

SUMMARY:
The purpose of this study is to determine if an automated text message intervention is beneficial for homeless patients in reducing their hospital visits, increasing their primary care appointments, and help them increase medication adherence.

DETAILED DESCRIPTION:
Boston Healthcare for the Homeless Program (BHCHP) is the study site for this research. It is the largest freestanding health care for the homeless program in the country - it provides primary care, behavioral health, oral health care and other wrap-around services to 12,500 homeless individuals a year. BHCHP was recently awarded a two-year grant from the Massachusetts Health Policy Commission to demonstrate how intensive, coordinated case management can reduce costs of caring for homeless persons who are high utilizers of emergency department (ED) and inpatient care. The Social Determinants of Health Coordinated Care Hub for Homeless Adults project (hereafter the "Care Hub") will create capacity among 9 Boston organizations serving homeless residents to meet their needs in primary care, behavioral health, housing, and shelter. This will improve quality of life, health outcomes, and care efficiency for the organizations. The participating organizations, in addition to BHCHP, are Bay Cove Human Services, Boston Public Health Commission, Boston Rescue Mission, Casa Esperanza, Massachusetts Housing and Shelter Alliance, The New England Center and Home for Veterans, St. Francis House, Victory Programs Specifically the investigators anticipate that patients participating in the Care Hub will have reduced use of ED and inpatient care because they will be better linked to and retained in appropriate care such as outpatient, mental health, substance use disorder (SUD), preventive care, and respite care. Regular care will increase the appropriate management of chronic health conditions and reduce episodes of exacerbations of these conditions which often lead to ED and hospital care. The purpose of this study is to evaluate whether an a text messaging system of appointment reminders, along with medication taking messages, and text messages about mood will augment the effectiveness of the Care Hub program.

The investigators propose to pilot a cell phone-based outpatient care support and medication reminder system. The content will include appointment reminders and educational and motivational messages about the importance of going to all outpatient care visits and of taking medications. The investigators take a community-based participatory research approach to this study - both because it appropriately considers the needs of the target population (increasing the likelihood of success) and because it empowers a population that is often treated as if its members were powerless. The cell phone texting intervention will help patients stay engaged in care, adhere to their medications, and adopt and sustain behavior change. This will be accomplished by completing a series of objectives:

1. To develop a text messaging system designed for homeless patients which includes appointment reminders, medication taking reminders and motivation, and texts messages that allow participants to report their mood, all in support of chronic disease management. The system will be based on a health coaching model, and message content will be reviewed and edited by patients who are members of drafted by patient members of a BHCHP Community Innovation Panel (CIP).
2. To train Care Hub intervention patients (or refresh existing skills) in cell phone text messaging.
3. To test the text messaging system in a randomized pilot study with 60 patients, comparing outpatient, respite care, ED, and inpatient utilization, and Health-Related Quality of Care (HRQOL) between the 30 intervention and 30 control patients.

ELIGIBILITY:
Inclusion Criteria:

* is a patient participant in the Coordinated Care Hub Initiative
* is willing to receive text messages
* is able to understand English - spoken and read

Exclusion Criteria:

* has an inability to find, open, and respond to a test text message

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Emergency Department Visits Made | 4 months
  Data from BHCHP's electronic medical record (EMR) and from the Coordinated Care Hub electronic case management system in use by the Care Hub organizations, which includes admission and discharge data

SECONDARY OUTCOMES:
Inpatient admissions | 4 months
  Similar to Emergency Department visit data, this will come from BHCHP's EMR and from the electronic case management system
Appointment keeping | 4 months
  Ratio of kept appointments to all appointments scheduled, based on the BHCHP EMR (e.g. 0-100%).
Medication Adherence | 4 months
  Self report medication adherence is assessed with 2 measures: Morisky adherence scale, (range, 0=poor to 11=excellent) and a 1-item rating question in which patients rate their ability to take all their medications as prescribed (range, 1=very poor to 6=excellent)
Adult Well-Being Assessment | 4 months
  This 9-item health-related quality of life (HRQOL) assessment is a validated measure developed by the Institute for Healthcare Improvement.
Comfort with Computers and Cell Phones | 4 months
  The eHealth Literacy Scale, eHEALS, (range 8-40, higher equals greater self-efficacy) assesses comfort with computers and the Internet for health related purposes. Investigators will also adapt eHEALS so that separate items can be asked about comfort with cell phone use.
Frequency of Cell Phone Use and Computer Use | 4 months
  Measures come from the Health Information National Trends Survey (HINTS). Scale ranges from 0 (no use) to 12 (frequent use of many features).
Outpatient appointments | 4 months
  Number of outpatient visits made

CONTACTS AND LOCATIONS:
Overall Officials: Donald K McInnes, ScD, Principal Investigator — Boston University and Department of Veterans Affairs
Locations (1):
- Boston University School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrow SM, Herman DB, Cordova P, Struening EL. Mortality among homeless shelter residents in New York City. Am J Public Health. 1999 Apr;89(4):529-34. doi: 10.2105/ajph.89.4.529. PMID 10191796
- [Background] Hwang SW, Aubry T, Palepu A, Farrell S, Nisenbaum R, Hubley AM, Klodawsky F, Gogosis E, Hay E, Pidlubny S, Dowbor T, Chambers C. The health and housing in transition study: a longitudinal study of the health of homeless and vulnerably housed adults in three Canadian cities. Int J Public Health. 2011 Dec;56(6):609-23. doi: 10.1007/s00038-011-0283-3. Epub 2011 Aug 20. PMID 21858461
- [Background] Krousel-Wood M, Thomas S, Muntner P, Morisky D. Medication adherence: a key factor in achieving blood pressure control and good clinical outcomes in hypertensive patients. Curr Opin Cardiol. 2004 Jul;19(4):357-62. doi: 10.1097/01.hco.0000126978.03828.9e. PMID 15218396
- [Background] Kidder DP, Wolitski RJ, Campsmith ML, Nakamura GV. Health status, health care use, medication use, and medication adherence among homeless and housed people living with HIV/AIDS. Am J Public Health. 2007 Dec;97(12):2238-45. doi: 10.2105/AJPH.2006.090209. Epub 2007 Oct 30. PMID 17971562
- [Background] Craig GM, Booth H, Story A, Hayward A, Hall J, Goodburn A, Zumla A. The impact of social factors on tuberculosis management. J Adv Nurs. 2007 Jun;58(5):418-24. doi: 10.1111/j.1365-2648.2007.04257.x. Epub 2007 Apr 17. PMID 17442025
- [Background] Kushel MB, Vittinghoff E, Haas JS. Factors associated with the health care utilization of homeless persons. JAMA. 2001 Jan 10;285(2):200-6. doi: 10.1001/jama.285.2.200. PMID 11176814
- [Background] Kushel MB, Perry S, Bangsberg D, Clark R, Moss AR. Emergency department use among the homeless and marginally housed: results from a community-based study. Am J Public Health. 2002 May;92(5):778-84. doi: 10.2105/ajph.92.5.778. PMID 11988447
- [Background] Clarke J, Proudfoot J, Ma H. Mobile Phone and Web-based Cognitive Behavior Therapy for Depressive Symptoms and Mental Health Comorbidities in People Living With Diabetes: Results of a Feasibility Study. JMIR Ment Health. 2016 May 31;3(2):e23. doi: 10.2196/mental.5131. PMID 27245948
- [Background] Nelson LA, Mulvaney SA, Gebretsadik T, Ho YX, Johnson KB, Osborn CY. Disparities in the use of a mHealth medication adherence promotion intervention for low-income adults with type 2 diabetes. J Am Med Inform Assoc. 2016 Jan;23(1):12-8. doi: 10.1093/jamia/ocv082. Epub 2015 Jul 17. PMID 26186935
- [Background] Whynes DK, MLitt BA, Giggs JA. The health of the Nottingham homeless. Public Health. 1992 Jul;106(4):307-14. doi: 10.1016/s0033-3506(05)80424-x. PMID 1529093
- [Background] Riley ED, Neilands TB, Moore K, Cohen J, Bangsberg DR, Havlir D. Social, structural and behavioral determinants of overall health status in a cohort of homeless and unstably housed HIV-infected men. PLoS One. 2012;7(4):e35207. doi: 10.1371/journal.pone.0035207. Epub 2012 Apr 25. PMID 22558128
- [Background] Emeche U. Is a strategy focused on super-utilizers equal to the task of health care system transformation? Yes. Ann Fam Med. 2015 Jan-Feb;13(1):6-7. doi: 10.1370/afm.1746. No abstract available. PMID 25583884
- [Background] Chambers C, Chiu S, Katic M, Kiss A, Redelmeier DA, Levinson W, Hwang SW. High utilizers of emergency health services in a population-based cohort of homeless adults. Am J Public Health. 2013 Dec;103 Suppl 2(Suppl 2):S302-10. doi: 10.2105/AJPH.2013.301397. Epub 2013 Oct 22. PMID 24148033
- [Background] Israel BA, Schulz AJ, Parker EA, Becker AB. Review of community-based research: assessing partnership approaches to improve public health. Annu Rev Public Health. 1998;19:173-202. doi: 10.1146/annurev.publhealth.19.1.173. PMID 9611617
- [Background] Larimer ME, Malone DK, Garner MD, Atkins DC, Burlingham B, Lonczak HS, Tanzer K, Ginzler J, Clifasefi SL, Hobson WG, Marlatt GA. Health care and public service use and costs before and after provision of housing for chronically homeless persons with severe alcohol problems. JAMA. 2009 Apr 1;301(13):1349-57. doi: 10.1001/jama.2009.414. PMID 19336710
- [Background] Mares AS, Rosenheck RA. Perceived relationship between military service and homelessness among homeless veterans with mental illness. J Nerv Ment Dis. 2004 Oct;192(10):715-9. doi: 10.1097/01.nmd.0000142022.08830.f4. PMID 15457118
- [Background] Mogollon-Pasapera E, Otvos L Jr, Giordano A, Cassone M. Bartonella: emerging pathogen or emerging awareness? Int J Infect Dis. 2009 Jan;13(1):3-8. doi: 10.1016/j.ijid.2008.04.002. Epub 2008 Jul 14. PMID 18621561
- [Background] Berg KM, Wilson IB, Li X, Arnsten JH. Comparison of antiretroviral adherence questions. AIDS Behav. 2012 Feb;16(2):461-8. doi: 10.1007/s10461-010-9864-z. PMID 21181252
- [Background] Lee SS, August GJ, Gewirtz AH, Klimes-Dougan B, Bloomquist ML, Realmuto GM. Identifying unmet mental health needs in children of formerly homeless mothers living in a supportive housing community sector of care. J Abnorm Child Psychol. 2010 Apr;38(3):421-32. doi: 10.1007/s10802-009-9378-1. PMID 20049523
- [Background] van der Vaart R, Drossaert CH, de Heus M, Taal E, van de Laar MA. Measuring actual eHealth literacy among patients with rheumatic diseases: a qualitative analysis of problems encountered using Health 1.0 and Health 2.0 applications. J Med Internet Res. 2013 Feb 11;15(2):e27. doi: 10.2196/jmir.2428. PMID 23399720
- [Background] van der Vaart R, van Deursen AJ, Drossaert CH, Taal E, van Dijk JA, van de Laar MA. Does the eHealth Literacy Scale (eHEALS) measure what it intends to measure? Validation of a Dutch version of the eHEALS in two adult populations. J Med Internet Res. 2011 Nov 9;13(4):e86. doi: 10.2196/jmir.1840. PMID 22071338
- [Background] Nelson DE, Kreps GL, Hesse BW, Croyle RT, Willis G, Arora NK, Rimer BK, Viswanath KV, Weinstein N, Alden S. The Health Information National Trends Survey (HINTS): development, design, and dissemination. J Health Commun. 2004 Sep-Oct;9(5):443-60; discussion 81-4. doi: 10.1080/10810730490504233. PMID 15513791
- [Background] Arora NK, Hesse BW, Rimer BK, Viswanath K, Clayman ML, Croyle RT. Frustrated and confused: the American public rates its cancer-related information-seeking experiences. J Gen Intern Med. 2008 Mar;23(3):223-8. doi: 10.1007/s11606-007-0406-y. Epub 2007 Oct 6. PMID 17922166
- [Background] Ivey SL, Tseng W, Kurtovich E, Lui B, Weir RC, Liu J, Song H, Wang M, Hubbard A. Evaluating a Culturally Competent Health Coach Intervention for Chinese American Patients with Diabetes. Diabetes Spectr. 2012 May 1;25(2):10.2337/diaspect.25.2.93. doi: 10.2337/diaspect.25.2.93. No abstract available. PMID 24311938